CLINICAL TRIAL: NCT01885507
Title: Duration of Mechanical Ventilation and Mortality Among Brain-injured Patients - a Before-after Evaluation of a Quality Improvement Project
Brief Title: Mechanical Ventilation in Brain-injured Patients
Acronym: BI-VILI
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC13_0127
Record Dates: First submitted 2013-06-18; First posted 2013-06-25 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-01

CONDITIONS: Brain-injury; Stroke; Subarachnoid Haemorrhage; Traumatic Brain Injury; Structural Coma
MeSH Terms: conditions — Brain Injuries; Stroke; Subarachnoid Hemorrhage; Brain Injuries, Traumatic | interventions — Airway Extubation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control phase (before): Process of care and outcomes before the educational program
- Training phase (after): Process of care and outcomes after the educational program which recommends:
  * the use of tidal volume < 7 ml/kg and of a positive expiratory pressure = 6 to 8 cmH20 (centimeter of water)
  * extubation as soon as ventilatory weaning is associated with a glasgow coma scale equal or above 10 and cough
  Interventions: Other: Pass recommendations on ventilation factors and extubation

INTERVENTIONS:
Other: Pass recommendations on ventilation factors and extubation — * the use of tidal volume < 7 ml/kg and of a positive expiratory pressure = 6 to 8 cmH20 (centimeter of water)
  * extubation as soon as ventilatory weaning is associated with a glasgow coma scale equal or above 10 and cough
  Groups: Training phase (after)

SUMMARY:
Protective ventilation (association of a tidal volume < 8 ml/kg with a positive end expiratory pressure) is poorly used in severe brain-injured patients. Moreover, a systematic approach to extubation may decrease the rate of extubation failure and enhance outcomes of brain-injured patients.

We hypothesized that medical education and implementation of an evidence-base care bundle associating protective ventilation and systemic approach to extubation can reduce the duration of mechanical ventilation in brain-injured patients.

DETAILED DESCRIPTION:
A before/after study design will be used. The before period (control phase) will consisted of all consecutive patients with severe brain-injury who were admitted to the participating ICUs.

During the interphase, all physicians, residents, physiotherapists and nurses will receive a formal training for the processes and procedures related to the 2 point bundle: protective ventilation and systematic approach to extubation (according to recommendation for the use of tidal volume < 7 ml/kg and of a positive expiratory pressure = 6 to 8 cmH20 (centimeter of water) and extubation as soon as ventilatory weaning is associated with a glasgow coma scale equal or above 10 and cought).

The after period consisted of all consecutive severe brain-injured patients admitted to the participating ICUs after the formal training.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (traumatic brain-injured, subarachnoid hemorrhage, stroke or other)
* Brain injury (Glasgow Coma Scale ≤ 12 associated with at least one anomaly related to an acute process on head tomographic tomodensitometry
* mechanical ventilation for more than 24 hours

Exclusion Criteria:

* early decision to withdraw care (taken in the first 24 hours in ICU),
* death in the first 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Structural coma.
Sampling Method: Non-Probability Sample
Enrollment: 560 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Mechanical ventilatory free days | Day-90
  The number of ventilator-free days was defined as the number of days from day 1 to day 90 on which a patient breaths spontaneously and is alive

SECONDARY OUTCOMES:
Mortality | day-90
In-ICU mortality | 90 days
Duration of mechanical ventilation | 90 days
ICU free days at day 90 | day 90
  The number of ICU free days was defined as the number of days from day 1 to on which a patient is alive and not hospitalized in ICU
Acute respiratory distress syndrome / acute lung injury | day-90
Hospital acquired pneumonia | day-90
Blood gaz | day-5
  PaO2 (arterial pressure of oxygen) and PaCO2 (arterial pressure of dioxide of carbon)
Intracranial pressure | day-5
Glasgow outcome scale | day-90
Extubation failure | day-90
Ventilatory setting | day-5
  Tidal volume and Positive end expiratory pressure

CONTACTS AND LOCATIONS:
Overall Officials: Karim Asehnoune, MD, PhD, Principal Investigator — Nantes University Hospital
Locations (22):
- France (22):
  - Angers University Hospital, Angers
  - Beaujon Hospital, Beaujon
  - Brest University Hospital, Brest
  - Caen University Hospital, Caen
  - Clermont-Ferrand University Hospital, Clermont-Ferrand
  - Henri Mondor University Hospital, Créteil
  - Grenoble University Hospital, Grenoble
  - Bicêtre University Hospital, Le Kremlin-Bicêtre
  - Marseille University Hospital, Marseille
  - Montpellier University Hospital, Montpellier
  - Nantes University Hospital, Nantes
  - Nice University Hospital, Nice
  - Nimes University Hospital, Nîmes
  - Georges Pompidou European Hospital, Paris
  - Poitiers University Hospital, Poitiers
  - Rennes University Hospital, Rennes
  - Rouen University Hospital, Rouen
  - Nantes University Hospital, Saint-Herblain
  - Toulouse University Hospital - Purpan, Toulouse
  - Toulouse University Hospital - Rangueil, Toulouse
  - Tours Univeristy Hospital - Neurosurgery ICU, Tours
  - Tours University Hospital - Neurotrauma ICU, Tours

REFERENCES:
- [Derived] Asehnoune K, Mrozek S, Perrigault PF, Seguin P, Dahyot-Fizelier C, Lasocki S, Pujol A, Martin M, Chabanne R, Muller L, Hanouz JL, Hammad E, Rozec B, Kerforne T, Ichai C, Cinotti R, Geeraerts T, Elaroussi D, Pelosi P, Jaber S, Dalichampt M, Feuillet F, Sebille V, Roquilly A; BI-VILI study group. A multi-faceted strategy to reduce ventilation-associated mortality in brain-injured patients. The BI-VILI project: a nationwide quality improvement project. Intensive Care Med. 2017 Jul;43(7):957-970. doi: 10.1007/s00134-017-4764-6. Epub 2017 Mar 18. PMID 28315940